CLINICAL TRIAL: NCT01589406
Title: Quality of Life and Sexuality in Women With Gynaecological Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 538-10CTIL
Record Dates: First submitted 2012-04-29; First posted 2012-05-02 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-04

CONDITIONS: Cancer
Keywords: Gynaecological Cancer; Quality of Life; Sexuality
MeSH Terms: conditions — Neoplasms; Sexuality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- group A group B: A:Patients for surgical intervention B:Patients for radiotherapy

SUMMARY:
Patients with premalignant (CIN3) and malignant cervical cancer will asked to complete questionnaires regarding intimacy (ENRICH) and life adaptation (PAIS) before treatment (surgery or radiotherapy) and after completion of treatment in order to estimate the influence of disease and treatment on quality of life indices.

DETAILED DESCRIPTION:
no additional information. see above

ELIGIBILITY:
Inclusion Criteria:

* women with Gynaecological cancer intended to undergo chemotherapy or surgery

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with Gynaecological cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 2 years
  longitudinal describtion of quality of life during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Amnon Amit, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel